CLINICAL TRIAL: NCT06218355
Title: IMPACT: Improving Maternal Postpartum Access to Care Through Telemedicine
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elaine Duryea, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2023-0332; PCORI-MMM-2022C2-27680 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-12-21; First posted 2024-01-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Complication
Keywords: telemedicine; hypertension; wound infection; readmission; metritis; mastitis; maternal mortality; postpartum complications
MeSH Terms: conditions — Hypertension; Wound Infection; Mastitis; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Education (Active Comparator): Women enrolled in the intensive education care model participate in intensive in-person education as well as ongoing virtual education via the electronic health record web portal in the form of strategically timed "pushes" of relevant and digestible educational elements via a "Care Companion." These virtual education "pushes" will include "to do" list reminders to check vital signs and submit them for review to the care team. Positive reinforcement will be provided when tasks are completed.
  Interventions: Other: Intensive Education
- Enhanced Virtual Care (Active Comparator): Women in the enhanced virtual care model will receive scheduled telehealth visits on the platform of their choice - either via video or audio-only synchronous visits. Patients in the virtual care model will check vital signs with home devices during the telehealth visit and report them directly to the provider. This "pull" approach to data collection directly contrasts with the "push" approach of comparator #1.
  Interventions: Other: Enhanced Virtual Care

INTERVENTIONS:
Other: Intensive Education — Intervention will consist of virtual education and communication through scheduled push notifications
  Arms: Intensive Education
Other: Enhanced Virtual Care — Intervention will utilize a telehealth model consisting of "pull" approach of patient engagement.
  Arms: Enhanced Virtual Care

SUMMARY:
The purpose of this study is to compare two complex, multi-component evidence-based postpartum interventions in underserved populations of lower socioeconomic status in an effort to reduce maternal morbidity and mortality.

DETAILED DESCRIPTION:
This large, multi-center randomized controlled trial will compare two multi-component postpartum care models via hybrid type 1 design conducted in two phases. An initial phase (phase 1) will collect baseline data and ensure patient input into final study. In phase 2, women will be randomized. Comparators are evidenced- based approaches: (1) an intensive in-person education with virtual education via push notifications using an electronic health record web portal; (2) a telehealth model using serial encounters. The "push" approach using notifications directly contrasts with the "pull" approach using telehealth visits. Both models include home visit programs. The study population includes patients delivering in two urban, inner-city health systems: Parkland (Dallas, TX) and Grady Memorial (Atlanta, GA). The primary outcome is time from hospital discharge to diagnosis and treatment of a composite of complications in the first 6 weeks. Based upon pilot data, 2349 women will demonstrate a 40% reduction (9 to 5.4 days) with 80% power and two-sided alpha of 0.05. 3500 women will be enrolled (1000 in phase 1; 2500 in phase 2) with anticipated <5% attrition at 6 weeks. Inclusion will be women who deliver liveborn infants. Secondary outcomes include mental health disorders, emergency room visits, hospital admissions, patient knowledge, quality of life and satisfaction, provider satisfaction, and social determinants of health. Women will be followed for one year postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who deliver a live born infant at Parkland Hospital or Grady Health and receive postpartum care at dedicated community clinics.
* Due to the nature of the study, all will be women, and all will be postpartum, thus of reproductive age. Postpartum women 18 years of age and older will be considered for inclusion if informed consent can be obtained.

Exclusion Criteria:

* Postpartum women who do not deliver at Parkland Hospital or Grady Health will not receive postpartum care in the pre-specified community clinics for Parkland health systems.
* Patients with a primary language other than English or Spanish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Healthcare Outcome - time to diagnosis and treatment of postpartum complications after hospital discharge | Up to one year postpartum
  Time to diagnosis and treatment of postpartum complications including hypertension, wound infection, and venous thromboembolism, measured in days. Lower value is considered better, representing timely care.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | enrollment, 1 week, 6 weeks, 3 months, 6 months, 1 year postpartum
  screening continuous, numerical; higher value consistent with great risk of postpartum depression
Generalized Anxiety Disorder 7 | enrollment, 1 week, 6 weeks, 3 months, 6 months, 1 year postpartum
  screening tool, continuous, numerical, higher value consistent with higher risk of anxiety disorder
Number of patients requiring emergency room visits, % preventable | Up to one year postpartum
  continuous variable, preventability to be determined by preventability panel
Number of patients requiring hospital admissions, % preventable | Up to one year postpartum
  continuous variable, preventability to be determined by preventability panel
Postpartum warning signs knowledge assessment, based on AWOHHN criteria | enrollment, 1 week, 6 weeks, 3 months, 6 months, 1 year postpartum
  Percent scored correct out of 10 total questions
PROMIS-29 questionnaire v 2.1 | 6 weeks and 1 year postpartum
  Scales 1-10 for each independent question, with numerical summary score
Healthy People 2030 questionnaire | 6 weeks and 1 year postpartum
  categorical variables selected by the participant
PRAPARE questionnaire | 6 weeks and 1 year postpartum
  categorical and dichotomous variables
Short Assessment of Patient Satisfaction (SAPS) | 6 weeks and 1 year postpartum
  Scale: Extremely dissatisfied to extremely satisfied Score Range is 0-28.
Provider Satisfaction Survey (Quantitative) | Every 6 months throughout the study period
  Scale: Strong agree to strongly disagree; very good to very bad; often to never
Systolic Blood Pressure | enrollment, 1 week, 6 weeks, 3 months, 6 months, 1 year postpartum
  numerical, continuous
Diastolic Blood Pressure | enrollment, 1 week, 6 weeks, 3 months, 6 months, 1 year postpartum
  numerical, continuous
Social Determinants of Health - Healthy People 2030 and PRAPARE questionnaire | enrollment, 6 weeks, 1 year postpartum
  qualitative data, each questions treated as dichotomous or categorical variables
Long-term disease control - diabetes - hemoglobin A1c, LDL, HDL, total cholesterol, triglycerides | enrollment, 6 weeks, 3 months, and 1 year postpartum
  laboratory value - continuous variables
Long-term disease control - hypertension - serum creatinine | enrollment, 6 weeks, 3 months, and 1 year postpartum
  laboratory value - continuous variable
Long-term disease control - liver function test (AST, ALT) | enrollment, 6 weeks, 3 months, and 1 year postpartum
  laboratory value - continuous variables
Long-term disease control - anemia - hemoglobin and hematocrit | enrollment, 6 weeks, 3 months, and 1 year postpartum
  laboratory value - continuous variables

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Duryea, MD, Principal Investigator — University of Texas Southwestern Medical Center; David B Nelson, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No